CLINICAL TRIAL: NCT06318390
Title: The Impact of KETO5 XOGenius Beverage on Markers of Physiological and Neurocognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Professor, The University of Texas at Arlington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0271
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Hypertension; Cognitive Decline; Diet; Healthy
Keywords: endothelial function; brain blood flow; cognition
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Keto5 XOGenius Beverage (Experimental): Keto5 XOGenius Beverage contains natural ingredients that are high in the Ketone β-OHB content and has anti-inflammatory and antioxidant properties
  Interventions: Dietary Supplement: XO Genius

INTERVENTIONS:
Dietary Supplement: XO Genius — This is a beverage powder that is high in healthy ingredients that are believed to be beneficial for physiological health

SUMMARY:
The primary objectives of this application are to 1) investigate the effect of increased daily consumption of the Keto5 XOGenius beverage on outcomes associated with elevated risk for various neurocognitive and pathophysiological conditions/diseases. And 2) to investigate the effect of daily consumption of the Keto5 XOGenius beverage on the following variables: waist circumference, body weight, and body mass index (BMI).

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality and affects all individuals. There are many primary risk factors for CVD with some of the primary causes including hypertension, hypercholesteremia, atherosclerosis, and type 2 diabetes mellitus. Furthermore, the rise in the prevalence of various neurocognitive conditions and cerebral vascular diseases including cognitive dysfunction, dementia, stroke, and Alzheimer's disease requires additional attention from a research perspective. While the reasons contributing to CVD and neurocognitive complications/cerebral vascular diseases, is multifactorial, a common link is impaired vascular function.

A hallmark of impaired vascular function is elevated arterial stiffness and a decrease in the vasodilator capacity in the brain and periphery. Reduced vascular function, due to elevated oxidative stress and systemic inflammation is implicated as a primary contributing factor for these attenuated vasodilatory responses. Therefore, it is reasonable to speculate that an approach targeting these pathways could abolish or minimize this elevated risk. One such approach could be increased dietary consumption of a naturally based product that is high in the ketone β-hydroxybutyrate (β-OHB). Importantly, recent research has indicated that short-term dietary supplementation (i.e. up to 14 days) of β-OHB has many important physiological benefits including improvements in peripheral and cerebral vascular function as well as cognitive function. Furthermore, it has been demonstrated that these beneficial effects are due in part to reductions in systemic oxidative stress and inflammation. Furthermore, this approach of oral supplementation has been demonstrated to be safe and well tolerated in various populations. In this regard, the overall research objective of this proposal is to determine the acute and chronic impact of daily supplementation of a Keto5 XOGenius on indices of physiological and neurocognitive health. Specifically, the Keto5 XOGenius is the product that we are interested in investigating in this proposal

The following objectives/aims will be explored:

1. Primary Aim - The primary endpoint is the effect of increased daily consumption of the Keto5 XOGenius beverage on outcomes associated with elevated risk for various neurocognitive and pathophysiological conditions/diseases. These outcomes include cognitive function, central and peripheral arterial blood pressure, cerebral and peripheral blood vessel function/health, and blood biomarkers (e.g., indices of inflammation, oxidative stress, insulin resistance/diabetes risk, and lipid profile).
2. Secondary Aim - A secondary endpoint is the effect of daily consumption of the Keto5 XOGenius beverage on the following variables: waist circumference, body weight, and body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are between the ages of 18-50

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, then we may still opt to proceed with data collection.
* Food allergies
* Type I diabetes/Type II diabetes, and/or a history of hypoglycemia.
* History of irritable bowel syndrome or inflammatory bowel disease.
* Currently taking any medications that are designed to treat a cardiovascular or metabolic condition
* Pregnant women
* Breast feeding women
* Allergy to spandex/lycra/latex
* Anemia
* Use of prescription stimulants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  Flow medicated dilation of the brachial artery (% change)
Neurocognitive Function | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  Performance on the NIH Toolbox Cognitive battery
Peripheral systolic blood pressure | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  standard blood pressure measures (mmHg)
Plasma concentration of Total Cholesterol (Total-C) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  assessment of Total Cholesterol
Arterial stiffness | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  assessment of pulse wave velocity and pulse wave analysis
Peripheral diastolic blood pressure (diastolic) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  standard blood pressure measures (mmHg)
Peripheral mean blood pressure (mean) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  standard blood pressure measures (mmHg)
Plasma concentration of High Density Lipoprotein (HDL-C) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  assessment of High Density Lipoprotein (HDL-C)
Plasma concentration of Low Density Lipoprotein (LDL-C) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  assessment of Low Density Lipoprotein (LDL-C)
Plasma concentration of Very Low Density Lipoprotein (VLDL-C) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  assessment of Low Density Lipoprotein (VLDL-C)
Plasma concentration of Triglycerides (TG) | baseline, 2 weeks post daily consumption of Keto5 XOgenius, & 4 weeks of daily keto5 XOgenius consumption
  assessment of Triglycerides (TG)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- UT Arlington - Science and Engineering Innovation and Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share IPD data